CLINICAL TRIAL: NCT06948682
Title: Exploring the Relationship Between Occlusion and Degenerative TMJ Disorders: A Comparative Clinical Study
Acronym: TMJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Khalid University (Other)
Responsible Party: Principal Investigator, Sunil Kumar Vaddamanu, Assistant Professor, King Khalid University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECC#2024-08
Record Dates: First submitted 2025-04-15; First posted 2025-04-29 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Degenerative Joint Disease; TMD
Keywords: TMD; Occlusal therapy; Degenerative joint disease; Pain management; Biomechanical stress
MeSH Terms: conditions — Joint Diseases; Agnosia | interventions — Occlusal Splints

STUDY DESIGN:
Intervention Model Description: study involves three separate groups of participants receiving different interventions:
  Group 1: Occlusal treatment
  Group 2: Conventional therapy
  Group 3: Standard management (control)
  Each participant is assigned to one group only and continues in that group throughout the study. This design is characteristic of a parallel assignment, where participants in different groups receive different interventions simultaneously.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Occlusal Treatment Group (Experimental): Participants in this group will receive occlusal treatment, including bite correction procedures and the use of occlusal splints, for a duration of 6 months. Monthly follow-ups will be conducted to monitor progress and make adjustments as needed.
  Interventions: Device: Occlusal Splint and Bite Correction Therapy; Other: Routine TMJ Care (Medication Only)
- Conventional Treatment Group (Active Comparator): Participants in this group will receive conventional TMJ therapy, including physical therapy, lifestyle modification counseling, and anti-inflammatory medications. Treatment is administered over 6 months with monthly clinical evaluations.
  Interventions: Other: Conventional TMJ Therapy
- Standard Care Group (No Intervention): Participants in this group will receive routine TMJ care involving only analgesic or anti-inflammatory medication as needed. No occlusal or physical therapy will be provided. Follow-up is conducted monthly for 6 months to assess standard care outcomes.

INTERVENTIONS:
Device: Occlusal Splint and Bite Correction Therapy — Participants receive individualized occlusal therapy involving occlusal splint use and bite correction (if needed). The treatment is applied continuously over a 6-month period. Monthly follow-up visits are conducted to monitor symptoms, adjust therapy, and evaluate radiographic changes in the TMJ.
  Arms: Occlusal Treatment Group
Other: Conventional TMJ Therapy — Participants undergo a 6-month conventional management program including pain medication (NSAIDs), physical therapy (jaw exercises, hot/cold therapy), and lifestyle guidance (diet modifications, stress reduction). Monthly clinical evaluations assess functional improvement and symptom reduction.
  Arms: Conventional Treatment Group
Other: Routine TMJ Care (Medication Only) — Participants receive standard pharmacological management for TMJ disorders (e.g., NSAIDs or analgesics) with no occlusal or physical therapy interventions. Follow-up assessments occur monthly for 6 months to monitor symptom progression and response to minimal intervention.
  Arms: Occlusal Treatment Group

SUMMARY:
The study "Exploring the Relationship Between Occlusion and Degenerative TMJ Disorders: A Comparative Clinical Study" investigated the efficacy of occlusal therapy in managing degenerative temporomandibular joint (TMJ) disorders. Conducted over 6 months with 150 patients, it compared three groups: occlusal therapy (Group 1), conventional treatment (Group 2), and routine care (Group 3). Group 1 showed significant improvements, including a 65% pain reduction, 51% better jaw function, slower joint degeneration, 64% less muscle tension, 24% improved jaw mobility, and enhanced quality of life, outperforming the other groups. The findings support occlusal therapy's role in multidisciplinary TMJ management, though long-term studies are needed.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 65 years

Clinical diagnosis of moderate to severe degenerative temporomandibular joint (TMJ) disorder, confirmed by:

Radiographic evidence (e.g., cartilage thinning, joint space narrowing)

Symptoms such as jaw pain, restricted jaw movement, or muscle tension

Ability to provide written informed consent

No recent trauma to the TMJ or oral structures

Exclusion Criteria:

Diagnosed rheumatoid arthritis or other autoimmune joint conditions

Serious cardiovascular, neurological, or systemic disorders

Pregnant women

Patients with contraindications for orthodontic procedures or occlusal splint use

History of TMJ surgery

Uncontrolled bruxism or other parafunctional habits that require alternative treatment strategies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-04-12 (Actual); Study Completion 2025-04-12 (Actual)

PRIMARY OUTCOMES:
Change in TMJ Pain Intensity (VAS Score) | Baseline, 3 months, and 6 months
  Assessment of temporomandibular joint pain using the Visual Analog Scale (VAS), scored from 0 (no pain) to 10 (worst possible pain). This outcome evaluates the effectiveness of occlusal treatment in reducing TMJ-related pain.
Change in Jaw Function (Jaw Function Limitation Scale - JFLS) | Baseline, 3 months, and 6 months
  Measurement of jaw functionality using the JFLS, a patient-reported scale ranging from 0 (no limitation) to 20 (severe limitation). This assesses improvements in jaw movement and function following different interventions.
Radiographic Changes in TMJ Structure | Baseline, 3 months, and 6 months
  Evaluation of TMJ degeneration using radiographic imaging (X-ray and MRI), including assessment of joint space narrowing, cartilage thinning, and subchondral bone changes. Quantitative imaging will compare structural changes across groups.

CONTACTS AND LOCATIONS:
Locations (1):
- King Khalid University, Abhā, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to confidentiality concerns and institutional policies restricting the distribution of patient-level data. While aggregated data may be published in scientific reports, raw individual-level data will remain confidential to protect participant privacy.